CLINICAL TRIAL: NCT01748643
Title: Effect of Deep Curarisation and Reversal With Sugammadex on Surgical Conditions and Perioperative Morbidity in Patients Undergoing Laparoscopic Gastric Bypass Surgery
Brief Title: CURES: The Effect of Deep Curarisation and Reversal With Sugammadex on Surgical Conditions and Perioperative Morbidity
Acronym: CURES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Pascal Vanelderen, M.D., Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PVRA-01; 2012-005533-37 (EudraCT Number); 8616-085MISP (Other Grant/Funding Number: MISP)
Record Dates: First submitted 2012-12-06; First posted 2012-12-12 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Laparoscopic Gastric Bypass Surgery; Surgical Conditions; Respiratory Function; Cerebral Tissue Oxygenation
MeSH Terms: conditions — Obesity; Respiratory Aspiration | interventions — Rocuronium; Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep neuromuscular blockade, reversal with sugammadex (Experimental): a continuous rocuronium infusion (0.6mg/kg (lean body mass)/h,) is started and titrated to a post tetanic count of 1-2 twitches. At the end of surgery neuromuscular blockade will be reversed with Sugammadex 4mg/kg. Patients are extubated when the train of four ratio is > 0.9.
  Interventions: Drug: deep neuromuscular blockade with rocuronium, reversal with sugammadex
- normal neuromuscular blockade, reversal with neostigmine (Active Comparator): After induction of anesthesia, top-ups of rocuronium (10mg) are given as needed to maintain a train of four count of 1-2. At the end of surgery neuromuscular blockade will be reversed with neostigmine 50μg/kg and glycopyrrolate 10μg/kg (lean body mass). Patients are extubated when TOF ratio > 0.9.
  Interventions: Drug: normal neuromuscular blockade reversal with rocuronium, reversal with neostigmine

INTERVENTIONS:
Drug: deep neuromuscular blockade with rocuronium, reversal with sugammadex — after induction of anesthesia, a rocuronium infusion (0.6mg/kg (lean body mass)/h,) is started and titrated to a post tetanic count of 1-2 twitches. At the end of surgery neuromuscular blockade will be reversed with sugammadex 4mg/kg. Patients are extubated when TOF ratio > 0.9.
  Other Names: rocuronium: Esmeron; sugammadex: Bridion
  Arms: Deep neuromuscular blockade, reversal with sugammadex
Drug: normal neuromuscular blockade reversal with rocuronium, reversal with neostigmine — After induction of anesthesia, top-ups of rocuronium (10mg) are given as needed to maintain a train of four count of 1-2. At the end of surgery neuromuscular blockade will be reversed with neostigmine 50μg/kg and glycopyrrolate 10μg/kg (lean body mass). Patients are extubated when the train of four ratio is > 0.9.
  Other Names: rocuronium: Esmeron; neostigmine; glycopyrrolate
  Arms: normal neuromuscular blockade, reversal with neostigmine

SUMMARY:
The purpose of this study is to investigate if a deep neuromuscular block with a continuous infusion of rocuronium titrated to a post-tetanic count (PTC) of 1-2 responses combined with reversal of neuromuscular blockade with sugammadex results in improved surgical conditions for the surgeon and/or improved post-operative respiratory function for the patients as compared to a standard technique with an intubation dose of rocuronium and top-ups as needed to maintain a neuromuscular blockade with a train of four (TOF) count of 1-2 and reversal of neuromuscular blockade with neostigmine/glycopyrrolate.

Furthermore, we want to investigate the effect of pneumoperitoneum, and NMB with rocuronium and reversal with sugammadex or neostigmine/glycopyrrolate on cerebral tissue oxygenation.

DETAILED DESCRIPTION:
Laparoscopic bariatric surgery poses special demands on the anaesthesiologist as well as the surgeon. The surgeon requires good visualisation of the operative field while the anaesthesiologist is concerned with adequate postoperative respiratory function in these morbidly obese patients. With the advent of advanced laparoscopic techniques the time span between adequate neuromuscular blockade (NMB) and adequate postoperative recovery of respiratory muscle function is growing ever shorter with an increasing risk of postoperative residual NMB.

Even minimal postoperative residual NMB with a train of four ratio (TOF) of 0.8 is associated with impaired respiratory function as witnessed in reductions of forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) in healthy volunteers. Moreover, a TOF < 0.7 correlates with increased postoperative respiratory complications due to the inability to swallow normally leading to aspiration, atelectasis and pneumonia. However, neuromuscular blocking agents not only impair respiratory function due to skeletal muscle relaxation. Also the body's response to hypoxia is impeded due to carotid body chemoreceptor suppression. Worryingly, reversal of NMB with neostigmine can lead to respiratory complications such as bronchospasm and even induce neuromuscular transmission failure in patients who already recovered from NMB.

Obese patients are at even greater risk for postoperative respiratory complications. In a recent study after bariatric surgery, 100% of patients had at least one hypoxic event (oxygen saturation <90% more then 30seconds). Restrictive ventilatory defects are clearly associated with body mass index (BMI) and obesity hypoventilation syndrome. Since respiratory failure is responsible for 11.8% of mortalities after bariatric surgery, optimal respiratory care for these patients is primordial. Optimal reversal of NMB plays an important role herein. With the advent of Sugammadex, a cyclodextrin molecule that encapsulates and inactivates rocuronium and vecuronium, rapid and dose-dependent reversal of profound NMB by high dose rocuronium is possible without the risk of impaired upper airway dilator muscle activity when given after recovery from NMB.

Furthermore, little is known about the cerebral tissue oxygen saturation (SctO2) in these morbidly obese patients during laparoscopic gastric bypass surgery. Since the unexpected finding that NMB influences hypoxic ventilatory response, more research is needed into the effect of neuromuscular blockers and their reversing agents on cerebral oxygenation. Using near infrared spectroscopy (Fore-sight®) technology absolute brain tissue oxygenation can be quantified to study these effects.

In this study we wish to investigate if a deep neuromuscular block with a continuous infusion of rocuronium titrated to a post-tetanic count (PTC) of 1-2 responses combined with reversal of NMB with sugammadex results in:

i. Improved surgical conditions for the surgeon ii. Improved post-operative respiratory function for the patients

as compared to a standard technique with an intubation dose of rocuronium and top-ups as needed to maintain a NMB with a TOF count of 1-2 and reversal of NMB with neostigmine/glycopyrrolate.

Furthermore, we wish to investigate the effect of pneumoperitoneum, and NMB with rocuronium and reversal with Sugammadex or neostigmine/glycopyrrolate on cerebral tissue oxygenation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent
2. American Society of Anaesthesiologists class I, II or III
3. Obese or morbid obese as defined by BMI > 30 and >40 kg/m2 respectively

Exclusion Criteria:

1. Neuromuscular disorders
2. Allergies to, or contraindication for muscle relaxants, neuromuscular reversing agents, anaesthetics, narcotics
3. Malignant hyperthermia
4. Pregnancy or lactation
5. Renal insufficiency defined as serum creatinine of 2x the upper normal limit, glomerular filtration rate < 60ml/min, urine output of < 0.5ml/kg/h for at least 6h
6. Chronic obstructive pulmonary disease GOLD classification 2 or higher.
7. Clinical, radiographic or laboratory findings suggesting upper or lower airway infection
8. Congestive heart failure.
9. Pickwick syndrome
10. Psychiatric illness inhibiting cooperation with study protocol or possibly obscuring results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter De Vooght, M.D., Study Chair — Ziekenhuis Oost-Limburg; Jeroen Van Melkebeek, M.D., Study Chair — Ziekenhuis Oost-Limburg; Dimitri Dylst, M.D., Study Chair — Ziekenhuis Oost-Limburg; Maud Beran, M.D., Study Chair — Ziekenhuis Oost-Limburg; Margot Vander Laenen, M.D., Study Chair — Ziekenhuis Oost-Limburg; Jan Van Zundert, M.D., PhD., Study Chair — Ziekenhuis Oost-Limburg; René Heylen, M.D., PhD., Study Chair — Ziekenhuis Oost-Limburg; Hans Verhelst, M.D., Study Chair — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Background] Ali HH, Wilson RS, Savarese JJ, Kitz RJ. The effect of tubocurarine on indirectly elicited train-of-four muscle response and respiratory measurements in humans. Br J Anaesth. 1975 May;47(5):570-4. doi: 10.1093/bja/47.5.570. PMID 1138775
- [Background] Eikermann M, Groeben H, Husing J, Peters J. Accelerometry of adductor pollicis muscle predicts recovery of respiratory function from neuromuscular blockade. Anesthesiology. 2003 Jun;98(6):1333-7. doi: 10.1097/00000542-200306000-00006. PMID 12766640
- [Background] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929
- [Background] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Eriksson LI. Reduced hypoxic chemosensitivity in partially paralysed man. A new property of muscle relaxants? Acta Anaesthesiol Scand. 1996 May;40(5):520-3. doi: 10.1111/j.1399-6576.1996.tb04482.x. PMID 8792879
- [Background] Wyon N, Joensen H, Yamamoto Y, Lindahl SG, Eriksson LI. Carotid body chemoreceptor function is impaired by vecuronium during hypoxia. Anesthesiology. 1998 Dec;89(6):1471-9. doi: 10.1097/00000542-199812000-00025. PMID 9856722
- [Background] Pratt CI. Bronchospasm after neostigmine. Anaesthesia. 1988 Mar;43(3):248. doi: 10.1111/j.1365-2044.1988.tb05560.x. No abstract available. PMID 3364648
- [Background] Payne JP, Hughes R, Al Azawi S. Neuromuscular blockade by neostigmine in anaesthetized man. Br J Anaesth. 1980 Jan;52(1):69-76. doi: 10.1093/bja/52.1.69. PMID 7378232
- [Background] Gallagher SF, Haines KL, Osterlund LG, Mullen M, Downs JB. Postoperative hypoxemia: common, undetected, and unsuspected after bariatric surgery. J Surg Res. 2010 Apr;159(2):622-6. doi: 10.1016/j.jss.2009.09.003. Epub 2009 Sep 25. PMID 20006346
- [Background] Saliman JA, Benditt JO, Flum DR, Oelschlager BK, Dellinger EP, Goss CH. Pulmonary function in the morbidly obese. Surg Obes Relat Dis. 2008 Sep-Oct;4(5):632-9; discussion 639. doi: 10.1016/j.soard.2008.06.010. Epub 2008 Jul 17. PMID 18722823
- [Background] Puhringer FK, Rex C, Sielenkamper AW, Claudius C, Larsen PB, Prins ME, Eikermann M, Khuenl-Brady KS. Reversal of profound, high-dose rocuronium-induced neuromuscular blockade by sugammadex at two different time points: an international, multicenter, randomized, dose-finding, safety assessor-blinded, phase II trial. Anesthesiology. 2008 Aug;109(2):188-97. doi: 10.1097/ALN.0b013e31817f5bc7. PMID 18648227
- [Background] Eikermann M, Zaremba S, Malhotra A, Jordan AS, Rosow C, Chamberlin NL. Neostigmine but not sugammadex impairs upper airway dilator muscle activity and breathing. Br J Anaesth. 2008 Sep;101(3):344-9. doi: 10.1093/bja/aen176. Epub 2008 Jun 16. PMID 18559352
- [Background] Cohen LB, Delegge MH, Aisenberg J, Brill JV, Inadomi JM, Kochman ML, Piorkowski JD Jr; AGA Institute. AGA Institute review of endoscopic sedation. Gastroenterology. 2007 Aug;133(2):675-701. doi: 10.1053/j.gastro.2007.06.002. No abstract available. PMID 17681185
- [Background] Miller MR, Dickinson SA, Hitchings DJ. The accuracy of portable peak flow meters. Thorax. 1992 Nov;47(11):904-9. doi: 10.1136/thx.47.11.904. PMID 1465746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13) | 42 (11) | 41.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 22 | 26 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 30 | 30 | 60
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 40 (3) | 41 (7) | 41 (5)
Peak expiratory flow [Mean (Standard Deviation); unit: L/min] | 314 (109) | 276 (81) | 295 (97)
Forced expiratory volume in 1 second [Mean (Standard Deviation); unit: L/min] | 2.4 (0.9) | 2.2 (0.6) | 2.3 (0.7)
Forced vital capacity [Mean (Standard Deviation); unit: L/min] | 3.0 (0.9) | 2.7 (0.8) | 2.8 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Evaluation of the View on the Operating Field by the Surgeon
Description: At the end of surgery, the view on the operating field will be graded by the surgeon using a 5-point rating scale:
  1. Extremely poor
  2. Poor
  3. Acceptable
  4. Good
  5. Optimal
Time Frame: Participants will be followed for the duration of the laparoscopic gastric bypass surgery, an expected average of 1.5h
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine
Number analyzed (Participants) | 30 | 30
units on a scale | 4.2 (1.0) | 3.9 (1.1)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade, Reversal With Sugammadex vs Normal Neuromuscular Blockade, Reversal With Neostigmine; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Intra-abdominal Pressure Rises > 18cmH2O
Description: The number of intra-abdominal pressure rises > 18cmH2O detected by the intra-abdominal CO2 insufflator.
Time Frame: Participants will be followed for the duration of the laparoscopic gastric bypass surgery, an expected average of 1.5h
Measure: Mean (Standard Deviation); unit: number of intra-abdominal pressure rises
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine
Number analyzed (Participants) | 30 | 30
number of intra-abdominal pressure rises | 0.2 (0.9) | 0.3 (1.0)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade, Reversal With Sugammadex vs Normal Neuromuscular Blockade, Reversal With Neostigmine; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Duration of Surgery
Description: Measured from the time of first skin incision to completion of skin closure.
Time Frame: Participants will be followed for the duration of the laparoscopic gastric bypass surgery, an expected average of 1.5h
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine
Number analyzed (Participants) | 30 | 30
minutes | 61.3 (15.1) | 70.6 (20.8)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade, Reversal With Sugammadex vs Normal Neuromuscular Blockade, Reversal With Neostigmine; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Peak Expiratory Flow
Description: Peak expiratory flow is measured with the Vitalograph® electronic portable peak flow meter. A mean of 3 measurements in the upright posture in bed before and after surgery will be used.
Time Frame: Measured the day before surgery and 30min after completion of surgery (when the modified observer's assessment of alertness/sedation scale is 5 (Patient responds readily to name spoken in normal tone))
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine
Number analyzed (Participants) | 30 | 30
percent change from baseline | 51.3 (31.6) | 51.5 (19.0)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade, Reversal With Sugammadex vs Normal Neuromuscular Blockade, Reversal With Neostigmine; Test type: Superiority; p = 0.97, t-test, 1 sided

5. Secondary Outcome: Forced Expiratory Volume in 1 Second
Description: Forced expiratory volume in 1 second is measured with the Vitalograph® electronic portable peak flow meter. A mean of 3 measurements in the upright posture in bed before and after surgery will be used.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine
Number analyzed (Participants) | 30 | 30
percent change from baseline | 45.2 (36.4) | 48.8 (19.6)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade, Reversal With Sugammadex vs Normal Neuromuscular Blockade, Reversal With Neostigmine; Test type: Superiority; p = 0.64, t-test, 1 sided

6. Secondary Outcome: Forced Vital Capacity
Description: Forced vital capacity is measured with the Vitalograph® electronic portable peak flow meter. A mean of 3 measurements in the upright posture in bed before and after surgery will be used.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine
Number analyzed (Participants) | 30 | 30
percent change from baseline | 51.9 (16.4) | 49.0 (22.6)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade, Reversal With Sugammadex vs Normal Neuromuscular Blockade, Reversal With Neostigmine; Test type: Superiority; p = 0.58, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Deep Neuromuscular Blockade, Reversal With Sugammadex | Normal Neuromuscular Blockade, Reversal With Neostigmine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No